CLINICAL TRIAL: NCT02741817
Title: WilL LOWer Dose Aspirin be More Effective Following ACS? (WILLOW-ACS)
Acronym: WILLOW-ACS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STH 19177
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2017-04

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin 20mg (Experimental): Supplied with sachets of 100mg soluble aspirin and training, instructions and equipment will be provided to prepare 20 mg dose twice daily x14 then aspirin 75mg once daily x14
  Interventions: Drug: Aspirin
- Aspirin 75mg (Experimental): This is the standard dose of aspirin the participant will already be taking. The study will require the participants to switch to soluble aspirin for two weeks to enable accurate comparison with the other dose and to take their aspirin dose in the morning. Participants will be provided with a supply of soluble aspirin, along with training, instructions and equipment to help prepare it. They should not take their usual aspirin tablets whilst receiving the study medication, but should continue all other usual medications.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — The intervention has been described previously in both arms individually. Group A will receive 20mg of soluble Aspirin and group B with 75mg of soluble Aspirin. As this is a crossover study, all patients will fall under both groups throughout the duration and be un-blinded.

SUMMARY:
The study is going to compare two different doses of aspirin for the treatment of heart disease in combination with the anticlotting medication ticagrelor. One of these doses of aspirin, 75 milligrams (mg) once a day, is the current standard treatment dose of aspirin used to treat heart attacks and angina. The other, 20 mg twice a day, is lower than the standard but there is growing scientific evidence that, when given with ticagrelor, this might offer advantages over the usual dose.

DETAILED DESCRIPTION:
Aspirin has an established role in the treatment of ACS and secondary prevention of ischaemic heart disease. In the landmark trial of aspirin in ACS, ISIS-2 (1988), it conferred a benefit of similar magnitude to thrombolysis. The addition of a second antiplatelet agent (a P2Y12 inhibitor) to aspirin is known to improve outcomes in both NSTE-ACS (Yusuf, Zhao et al. 2001) and STEMI (Chen, Jiang et al. 2005, Sabatine, Cannon et al. 2005). There are 2 major classes of oral P2Y12 inhibitor: irreversibly binding thienopyridine agents, such as clopidogrel or prasugrel, and reversibly-binding drugs, such as the cyclo-pentyl triazolopyrimidine ticagrelor.

A combination of aspirin and ticagrelor 90 milligrams (mg) twice daily for at least 1 year represents the current standard treatment for ACS recommended in European guidelines (Steg, James et al. 2012, Roffi, Patrono et al. 2015).

Aspirin inhibits cyclo-oxygenase (COX) enzymes by irreversible acetylation, and at lower doses exhibits relative selectivity for COX1, responsible for the synthesis of thromboxane A2 (TXA2), which is a pro-thrombotic and vasoconstrictive eicosanoid. At higher doses, aspirin is also able to inhibit COX2, leading to a reduction in release of the anti-thrombotic and vasodilatory compound prostacyclin (PGI2). Aspirin is able to inhibit platelet aggregation, therefore, by inhibiting TXA2 relatively more than PGI2. Due to its irreversible binding, COX is inhibited in platelets for their lifespan (typically 10-12 days) as, being without a nucleus, they cannot regenerate the enzyme (Patrono 1994). It is now thought that PGI2 acts locally rather than systemically and, in healthy individuals, COX1 may be responsible for the majority of PGI2 production (Kirkby, Lundberg et al. 2012). In patients with atheromatous disease, however, there is greater COX2 expression in diseased vessel walls (Schonbeck, Sukhova et al. 1999) therefore this may not apply in the areas most vulnerable to thrombosis. COX2 selective inhibitors have been associated with increased cardiovascular risk and this appears to be both a dose dependent and class effect (Mukherjee, Nissen et al. 2001, Bhala, Emberson et al. 2013).

All antithrombotic drugs confer a risk of bleeding. In addition to its antiplatelet effect, COX1 inhibition by aspirin in the stomach can lead to acid-induced inflammation and ulceration, resulting in bleeding. There is evidence that lower doses of aspirin are associated with lower rates of gastrointestinal bleeding (Valkhoff, Sturkenboom et al. 2012) including when combined with a P2Y12 inhibitor (Mehta, Tanguay et al. 2010).

In the UK, 75 mg od is the standard maintenance dose of aspirin and the consensus from the Antithrombotic Trialist Collaborators was that higher doses offer no added benefit and may increase complication rates when used for secondary prevention (2002). Use of this specific dose stems from its original formulation as an anti-inflammatory dose for paediatric use, and was chosen to approximate 1 grain in the formerly used unit. Only 1 study of aspirin dose in patients with ACS on DAPT has been carried out but this only included patients on clopidogrel rather than ticagrelor and did not evaluate aspirin doses lower than 75 mg (Mehta, Tanguay et al. 2010).

Aspirin and ticagrelor are superior to aspirin and clopidogrel in preventing ischaemic complications in ACS but there is an increased rate of bleeding complications (Wallentin, Becker et al. 2009). There is some evidence that the benefit of ticagrelor over clopidogrel was diminished in patients taking higher doses of aspirin compared to lower doses (Mahaffey, Wojdyla et al. 2011).

The P2Y12 and arachidonic acid pathways appear to be linked. P2Y12 inhibition has been shown to reduce TXA2 release from platelets (Armstrong, Leadbeater et al. 2011) and potentiates the antiplatelet effect of PGI2 in vitro (Cattaneo and Lecchi 2007). Ticagrelor acts as a more potent P2Y12 inhibitor than clopidogrel (Storey, Angiolillo et al. 2010) and therefore may contribute more to this.

Ticagrelor has pleiotropic effects not seen with clopidogrel, including inhibition of erythrocyte adenosine uptake (Bonello, Laine et al. 2014) and, in a preclinical model, reduction of infarct size, an adenosine and COX2 dependent effect that is inhibited by high but not low dose aspirin (Nanhwan, Ling et al. 2014). Chronic, but not acute, ticagrelor treatment may upregulate COX2 expression (Nanhwan, Ling et al. 2014) and ticagrelor, but not clopidogrel, improves post-infarct remodeling (Ye, Birnbaum et al. 2015) and has an anticontractile effect on vascular smooth muscle cells when exposed to ADP which is inhibited by high dose, but not low dose, aspirin (Grzesk, Kozinski et al. 2013).

Additionally, statins, given to the majority of patients with ACS, reduce infarct size by a COX2 dependent mechanism and, again, this effect is inhibited by aspirin in a dose-dependent manner (Birnbaum, Lin et al. 2007). Inhibition of COX2 by higher doses of aspirin therefore may reduce these benefits.

In healthy volunteer studies, aspirin at a dose of 75 mg once daily provided only a small additional effect on platelets to prasugrel ex vivo (Leadbeater et al 2011) and similar findings have been shown with prasugrel (Armstrong et al 2011) and ticagrelor (Kirkby et al 2011) in vitro, however the clinical significance of this additional effect is not known as studies have not been made in patients with acute coronary syndrome, in whom platelet activation occurs and persists after the acute period (Ault, Cannon et al. 1999).

It has been suggested that ticagrelor monotherapy may in fact offer advantages over DAPT (Warner, Armstrong et al. 2010) and 2 trials including ACS patients after the very early period are currently in progress (National Institutes of Health 2014, National Institutes of Health 2015). However, given the fact that aspirin still possesses some antiplatelet effect in the presence of potent P2Y12 inhibition, its total omission may not prove to be the optimum strategy in higher risk patients, particularly given the current lack of evidence in patients rather than healthy individuals.

Aspirin inhibits TXA2 and PGI2 in vivo in a dose dependent manner and daily doses as low as 20 mg have been shown to significantly inhibit TXA2 release (Warner, Nylander et al. 2011), whilst similar doses provide minimal PGI2 inhibition and no significant prolongation of the bleeding time (Kallmann, Nieuwenhuis et al. 1987). Aspirin doses of less than 75mg OD have not been studied in combination with P2Y12 inhibitors. A strategy to reduce the effect of aspirin on beneficial COX2 whilst maintaining its antiplatelet effect in the presence of ticagrelor may therefore be a lower dose than the current standard.

Dosing frequency may also be open to optimization. Aspirin is cleared from the plasma quickly after administration but its effect lasts for the lifespan of a platelet due to its properties as an irreversible inhibitor (Patrono 1994). However, a significant proportion of the population have a high rate of platelet turnover that therefore reduces the duration of effect and may lead to inadequate platelet inhibition. This has been shown to be the case in patients with ischaemic heart disease and is most frequently a problem in those with diabetes mellitus, obesity and smokers (Henry, Vermillet et al. 2011). Twice-daily dosing may offer more consistency (Rocca, Santilli et al. 2012, Paikin, Hirsh et al. 2015). Again, this has not been studied when in combination with a P2Y12 inhibitor. As ticagrelor is taken twice daily, it would not significantly inconvenience patients to receive doses of aspirin in this way.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, subjects should fulfill the following criteria:

1. Provision of informed consent prior to any study specific procedures
2. Male or female aged greater than 18 years
3. Previous diagnosis of acute coronary syndrome greater than 30 days and less than 10 months before enrollment
4. Receiving dual antiplatelet therapy with aspirin 75 mg once daily and ticagrelor 90 mg twice daily

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Presence of an indication for dual antiplatelet therapy other than ischaemic heart disease
2. PCI with drug eluting or bare metal stent(s) within 30 days of randomization
3. Any history of stent implantation to the left main coronary artery
4. Any history of stent thrombosis during dual antiplatelet therapy
5. Planned procedure for coronary revascularization
6. Any planned surgery or other procedure that may require suspension or discontinuation of dual antiplatelet therapy expected to occur within 3 months of randomisation
7. Prior intention by patient or physician to discontinue aspirin and/or ticagrelor within the study period
8. Receiving doses of aspirin and ticagrelor other than 75 mg once daily and 90mg twice daily respectively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06-26 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
Post-dose serum thromboxane B2, compared within-patients between the 2 dosing regimens by a paired t test. | Approx 12 months from start date
Post-dose urinary PGI-M, compared within-patients between the 2 dosing regimens by a paired t test. | Approx 12 months from start date
Ratio of post-dose serum TXB2:urinary PGI-M, compared within-patients between the 2 dosing regimens by a paired t test. | Approx 12 months from start date

SECONDARY OUTCOMES:
Pre-dose serum thromboxane B2, compared within-patients between the 2 dosing regimens by a paired t test. | Approx 12 months from start date
Maximum and final post-dose platelet aggregation induced by 0.1, 0.3 and 1 mM arachidonic acid; 1, 4 and 16 µg/ml collagen; and 20 µM ADP compared within-patients between the 2 dosing regimens by paired t tests. | Approx 12 months from start date
Maximum and final pre-dose platelet aggregation induced by 0.1, 0.3 and 1 mM arachidonic acid; 1, 4 and 16 µg/ml collagen; and 20 µM ADP compared within-patients between the 2 dosing regimens by paired t tests. | Approx 12 months from start date
Post-dose bleeding time compared within-patients between the 2 dosing regimens by a paired t test. | Approx 12 months from start date
Ratio of pre-:post-dose serum TXB2, compared within-patients between the 2 dosing regimens by a paired t test. | Approx 12 months from start date
Ratio of pre-:post-dose maximum and final platelet aggregation induced by 0.1, 0.3 and 1 mM arachidonic acid; 1, 4 and 16 µg/ml collagen; and 20 µM ADP compared within-patients between the 2 dosing regimens by paired t tests. | Approx 12 months from start date

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Randomised trial of intravenous streptokinase, oral aspirin, both, or neither among 17,187 cases of suspected acute myocardial infarction: ISIS-2. ISIS-2 (Second International Study of Infarct Survival) Collaborative Group. Lancet. 1988 Aug 13;2(8607):349-60. PMID 2899772
- [Background] Antithrombotic Trialists' Collaboration. Collaborative meta-analysis of randomised trials of antiplatelet therapy for prevention of death, myocardial infarction, and stroke in high risk patients. BMJ. 2002 Jan 12;324(7329):71-86. doi: 10.1136/bmj.324.7329.71. PMID 11786451
- [Background] Armstrong PC, Leadbeater PD, Chan MV, Kirkby NS, Jakubowski JA, Mitchell JA, Warner TD. In the presence of strong P2Y12 receptor blockade, aspirin provides little additional inhibition of platelet aggregation. J Thromb Haemost. 2011 Mar;9(3):552-61. doi: 10.1111/j.1538-7836.2010.04160.x. PMID 21143373
- [Background] Ault KA, Cannon CP, Mitchell J, McCahan J, Tracy RP, Novotny WF, Reimann JD, Braunwald E. Platelet activation in patients after an acute coronary syndrome: results from the TIMI-12 trial. Thrombolysis in Myocardial Infarction. J Am Coll Cardiol. 1999 Mar;33(3):634-9. doi: 10.1016/s0735-1097(98)00635-4. PMID 10080462
- [Background] Coxib and traditional NSAID Trialists' (CNT) Collaboration; Bhala N, Emberson J, Merhi A, Abramson S, Arber N, Baron JA, Bombardier C, Cannon C, Farkouh ME, FitzGerald GA, Goss P, Halls H, Hawk E, Hawkey C, Hennekens C, Hochberg M, Holland LE, Kearney PM, Laine L, Lanas A, Lance P, Laupacis A, Oates J, Patrono C, Schnitzer TJ, Solomon S, Tugwell P, Wilson K, Wittes J, Baigent C. Vascular and upper gastrointestinal effects of non-steroidal anti-inflammatory drugs: meta-analyses of individual participant data from randomised trials. Lancet. 2013 Aug 31;382(9894):769-79. doi: 10.1016/S0140-6736(13)60900-9. Epub 2013 May 30. PMID 23726390
- [Background] Birnbaum Y, Lin Y, Ye Y, Martinez JD, Huang MH, Lui CY, Perez-Polo JR, Uretsky BF. Aspirin before reperfusion blunts the infarct size limiting effect of atorvastatin. Am J Physiol Heart Circ Physiol. 2007 Jun;292(6):H2891-7. doi: 10.1152/ajpheart.01269.2006. Epub 2007 Feb 2. PMID 17277020
- [Background] Bonello L, Laine M, Kipson N, Mancini J, Helal O, Fromonot J, Gariboldi V, Condo J, Thuny F, Frere C, Camoin-Jau L, Paganelli F, Dignat-George F, Guieu R. Ticagrelor increases adenosine plasma concentration in patients with an acute coronary syndrome. J Am Coll Cardiol. 2014 Mar 11;63(9):872-7. doi: 10.1016/j.jacc.2013.09.067. Epub 2013 Nov 27. PMID 24291273
- [Background] Cannon CP, Husted S, Harrington RA, Scirica BM, Emanuelsson H, Peters G, Storey RF; DISPERSE-2 Investigators. Safety, tolerability, and initial efficacy of AZD6140, the first reversible oral adenosine diphosphate receptor antagonist, compared with clopidogrel, in patients with non-ST-segment elevation acute coronary syndrome: primary results of the DISPERSE-2 trial. J Am Coll Cardiol. 2007 Nov 6;50(19):1844-51. doi: 10.1016/j.jacc.2007.07.053. Epub 2007 Oct 23. PMID 17980250
- [Background] Cattaneo M, Lecchi A. Inhibition of the platelet P2Y12 receptor for adenosine diphosphate potentiates the antiplatelet effect of prostacyclin. J Thromb Haemost. 2007 Mar;5(3):577-82. doi: 10.1111/j.1538-7836.2007.02356.x. Epub 2006 Dec 7. PMID 17155953
- [Background] Chen ZM, Jiang LX, Chen YP, Xie JX, Pan HC, Peto R, Collins R, Liu LS; COMMIT (ClOpidogrel and Metoprolol in Myocardial Infarction Trial) collaborative group. Addition of clopidogrel to aspirin in 45,852 patients with acute myocardial infarction: randomised placebo-controlled trial. Lancet. 2005 Nov 5;366(9497):1607-21. doi: 10.1016/S0140-6736(05)67660-X. PMID 16271642
- [Background] Favre L, Glasson P, Riondel A, Vallotton MB. Interaction of diuretics and non-steroidal anti-inflammatory drugs in man. Clin Sci (Lond). 1983 Apr;64(4):407-15. doi: 10.1042/cs0640407. PMID 6337769
- [Background] Grzesk G, Kozinski M, Tantry US, Wicinski M, Fabiszak T, Navarese EP, Grzesk E, Jeong YH, Gurbel PA, Kubica J. High-dose, but not low-dose, aspirin impairs anticontractile effect of ticagrelor following ADP stimulation in rat tail artery smooth muscle cells. Biomed Res Int. 2013;2013:928271. doi: 10.1155/2013/928271. Epub 2013 Jun 6. PMID 23841099
- [Background] Henry P, Vermillet A, Boval B, Guyetand C, Petroni T, Dillinger JG, Sideris G, Bal dit Sollier C, Drouet L. 24-hour time-dependent aspirin efficacy in patients with stable coronary artery disease. Thromb Haemost. 2011 Feb;105(2):336-44. doi: 10.1160/TH10-02-0082. Epub 2010 Dec 7. PMID 21136023
- [Background] Kallmann R, Nieuwenhuis HK, de Groot PG, van Gijn J, Sixma JJ. Effects of low doses of aspirin, 10 mg and 30 mg daily, on bleeding time, thromboxane production and 6-keto-PGF1 alpha excretion in healthy subjects. Thromb Res. 1987 Feb 15;45(4):355-61. doi: 10.1016/0049-3848(87)90224-6. PMID 3576521
- [Background] Kirkby NS, Lundberg MH, Harrington LS, Leadbeater PD, Milne GL, Potter CM, Al-Yamani M, Adeyemi O, Warner TD, Mitchell JA. Cyclooxygenase-1, not cyclooxygenase-2, is responsible for physiological production of prostacyclin in the cardiovascular system. Proc Natl Acad Sci U S A. 2012 Oct 23;109(43):17597-602. doi: 10.1073/pnas.1209192109. Epub 2012 Oct 8. PMID 23045674
- [Background] Mahaffey KW, Wojdyla DM, Carroll K, Becker RC, Storey RF, Angiolillo DJ, Held C, Cannon CP, James S, Pieper KS, Horrow J, Harrington RA, Wallentin L; PLATO Investigators. Ticagrelor compared with clopidogrel by geographic region in the Platelet Inhibition and Patient Outcomes (PLATO) trial. Circulation. 2011 Aug 2;124(5):544-54. doi: 10.1161/CIRCULATIONAHA.111.047498. Epub 2011 Jun 27. PMID 21709065
- [Background] Matetzky S, Shenkman B, Guetta V, Shechter M, Beinart R, Goldenberg I, Novikov I, Pres H, Savion N, Varon D, Hod H. Clopidogrel resistance is associated with increased risk of recurrent atherothrombotic events in patients with acute myocardial infarction. Circulation. 2004 Jun 29;109(25):3171-5. doi: 10.1161/01.CIR.0000130846.46168.03. Epub 2004 Jun 7. PMID 15184279
- [Background] Mehta SR, Tanguay JF, Eikelboom JW, Jolly SS, Joyner CD, Granger CB, Faxon DP, Rupprecht HJ, Budaj A, Avezum A, Widimsky P, Steg PG, Bassand JP, Montalescot G, Macaya C, Di Pasquale G, Niemela K, Ajani AE, White HD, Chrolavicius S, Gao P, Fox KA, Yusuf S; CURRENT-OASIS 7 trial investigators. Double-dose versus standard-dose clopidogrel and high-dose versus low-dose aspirin in individuals undergoing percutaneous coronary intervention for acute coronary syndromes (CURRENT-OASIS 7): a randomised factorial trial. Lancet. 2010 Oct 9;376(9748):1233-43. doi: 10.1016/S0140-6736(10)61088-4. PMID 20817281
- [Background] Miner J, Hoffhines A. The discovery of aspirin's antithrombotic effects. Tex Heart Inst J. 2007;34(2):179-86. PMID 17622365
- [Background] Mukherjee D, Nissen SE, Topol EJ. Risk of cardiovascular events associated with selective COX-2 inhibitors. JAMA. 2001 Aug 22-29;286(8):954-9. doi: 10.1001/jama.286.8.954. PMID 11509060
- [Background] Nanhwan MK, Ling S, Kodakandla M, Nylander S, Ye Y, Birnbaum Y. Chronic treatment with ticagrelor limits myocardial infarct size: an adenosine and cyclooxygenase-2-dependent effect. Arterioscler Thromb Vasc Biol. 2014 Sep;34(9):2078-85. doi: 10.1161/ATVBAHA.114.304002. Epub 2014 Jul 10. PMID 25012137
- [Background] Paikin JS, Hirsh J, Ginsberg JS, Weitz JI, Chan NC, Whitlock RP, Pare G, Johnston M, Eikelboom JW. Multiple daily doses of acetyl-salicylic acid (ASA) overcome reduced platelet response to once-daily ASA after coronary artery bypass graft surgery: a pilot randomized controlled trial. J Thromb Haemost. 2015 Mar;13(3):448-56. doi: 10.1111/jth.12832. Epub 2015 Feb 6. PMID 25546465
- [Background] Patrono C. Aspirin as an antiplatelet drug. N Engl J Med. 1994 May 5;330(18):1287-94. doi: 10.1056/NEJM199405053301808. No abstract available. PMID 8145785
- [Background] Pradelles P, Grassi J, Maclouf J. Enzyme immunoassays of eicosanoids using acetylcholinesterase. Methods Enzymol. 1990;187:24-34. doi: 10.1016/0076-6879(90)87005-n. No abstract available. PMID 2233347
- [Background] Rocca B, Santilli F, Pitocco D, Mucci L, Petrucci G, Vitacolonna E, Lattanzio S, Mattoscio D, Zaccardi F, Liani R, Vazzana N, Del Ponte A, Ferrante E, Martini F, Cardillo C, Morosetti R, Mirabella M, Ghirlanda G, Davi G, Patrono C. The recovery of platelet cyclooxygenase activity explains interindividual variability in responsiveness to low-dose aspirin in patients with and without diabetes. J Thromb Haemost. 2012 Jul;10(7):1220-30. doi: 10.1111/j.1538-7836.2012.04723.x. PMID 22471290
- [Background] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Background] Sabatine MS, Cannon CP, Gibson CM, Lopez-Sendon JL, Montalescot G, Theroux P, Claeys MJ, Cools F, Hill KA, Skene AM, McCabe CH, Braunwald E; CLARITY-TIMI 28 Investigators. Addition of clopidogrel to aspirin and fibrinolytic therapy for myocardial infarction with ST-segment elevation. N Engl J Med. 2005 Mar 24;352(12):1179-89. doi: 10.1056/NEJMoa050522. Epub 2005 Mar 9. PMID 15758000
- [Background] Schonbeck U, Sukhova GK, Graber P, Coulter S, Libby P. Augmented expression of cyclooxygenase-2 in human atherosclerotic lesions. Am J Pathol. 1999 Oct;155(4):1281-91. doi: 10.1016/S0002-9440(10)65230-3. PMID 10514410
- [Background] Task Force on the management of ST-segment elevation acute myocardial infarction of the European Society of Cardiology (ESC); Steg PG, James SK, Atar D, Badano LP, Blomstrom-Lundqvist C, Borger MA, Di Mario C, Dickstein K, Ducrocq G, Fernandez-Aviles F, Gershlick AH, Giannuzzi P, Halvorsen S, Huber K, Juni P, Kastrati A, Knuuti J, Lenzen MJ, Mahaffey KW, Valgimigli M, van 't Hof A, Widimsky P, Zahger D. ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Eur Heart J. 2012 Oct;33(20):2569-619. doi: 10.1093/eurheartj/ehs215. Epub 2012 Aug 24. No abstract available. PMID 22922416
- [Background] Storey RF, Angiolillo DJ, Patil SB, Desai B, Ecob R, Husted S, Emanuelsson H, Cannon CP, Becker RC, Wallentin L. Inhibitory effects of ticagrelor compared with clopidogrel on platelet function in patients with acute coronary syndromes: the PLATO (PLATelet inhibition and patient Outcomes) PLATELET substudy. J Am Coll Cardiol. 2010 Oct 26;56(18):1456-62. doi: 10.1016/j.jacc.2010.03.100. PMID 20832963
- [Background] Storey RF, Oldroyd KG, Wilcox RG. Open multicentre study of the P2T receptor antagonist AR-C69931MX assessing safety, tolerability and activity in patients with acute coronary syndromes. Thromb Haemost. 2001 Mar;85(3):401-7. PMID 11307804
- [Background] Tohgi H, Konno S, Tamura K, Kimura B, Kawano K. Effects of low-to-high doses of aspirin on platelet aggregability and metabolites of thromboxane A2 and prostacyclin. Stroke. 1992 Oct;23(10):1400-3. doi: 10.1161/01.str.23.10.1400. PMID 1412574
- [Background] Valkhoff VE, Sturkenboom MC, Kuipers EJ. Risk factors for gastrointestinal bleeding associated with low-dose aspirin. Best Pract Res Clin Gastroenterol. 2012 Apr;26(2):125-40. doi: 10.1016/j.bpg.2012.01.011. PMID 22542151
- [Background] Vane JR, Botting RM. The mechanism of action of aspirin. Thromb Res. 2003 Jun 15;110(5-6):255-8. doi: 10.1016/s0049-3848(03)00379-7. PMID 14592543
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Background] Warner TD, Armstrong PC, Curzen NP, Mitchell JA. Dual antiplatelet therapy in cardiovascular disease: does aspirin increase clinical risk in the presence of potent P2Y12 receptor antagonists? Heart. 2010 Nov;96(21):1693-4. doi: 10.1136/hrt.2010.205724. PMID 20956485
- [Background] Warner TD, Nylander S, Whatling C. Anti-platelet therapy: cyclo-oxygenase inhibition and the use of aspirin with particular regard to dual anti-platelet therapy. Br J Clin Pharmacol. 2011 Oct;72(4):619-33. doi: 10.1111/j.1365-2125.2011.03943.x. PMID 21320154
- [Background] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Background] Ye Y, Birnbaum GD, Perez-Polo JR, Nanhwan MK, Nylander S, Birnbaum Y. Ticagrelor protects the heart against reperfusion injury and improves remodeling after myocardial infarction. Arterioscler Thromb Vasc Biol. 2015 Aug;35(8):1805-14. doi: 10.1161/ATVBAHA.115.305655. Epub 2015 Jun 4. PMID 26044583
- [Background] Yusuf S, Zhao F, Mehta SR, Chrolavicius S, Tognoni G, Fox KK; Clopidogrel in Unstable Angina to Prevent Recurrent Events Trial Investigators. Effects of clopidogrel in addition to aspirin in patients with acute coronary syndromes without ST-segment elevation. N Engl J Med. 2001 Aug 16;345(7):494-502. doi: 10.1056/NEJMoa010746. PMID 11519503